CLINICAL TRIAL: NCT01185613
Title: Clinical Evaluation of Therapy™ Cool Flex Ablation Catheter for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: FACT-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Christophe Bailleul, SJM International, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AF-09-024-EU-AB
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapy™ Cool Flex Ablation Catheter (Experimental)
  Interventions: Device: Therapy™ Cool Flex Ablation Catheter

INTERVENTIONS:
Device: Therapy™ Cool Flex Ablation Catheter — The device under evaluation is the 4mm Therapy™ Cool Flex Ablation Catheter. The Therapy™ Cool Flex catheter is a flexible tip, insulated, 7F catheter constructed of thermoplastic elastomer material and noble metal electrodes.
  The following CE Mark devices will be used in conjunction with the Therapy™ Cool Flex Ablation Catheter
  * IBI-1500T11 Cardiac Ablation Generator (RF ablation generator) with software version 3.0 or higher.
  * Cool Point™ Irrigation Pump
  * Cool Point™ Tubing set
  * Data Logger

SUMMARY:
The purpose of this study is to observe the performance of Therapy™ Cool Flex™ catheter by documenting the procedural parameters, major complications and recurrence of AF after ablation using Cool Flex ablation catheter for the treatment of paroxysmal atrial fibrillation.

This study is an observational clinical study which is not based on any specific endpoints.

ELIGIBILITY:
Inclusion Criteria:

* A signed written Informed Consent form
* 18 years of age or older
* Agrees to comply with follow-up visits and evaluation
* Candidate for catheter ablation for the treatment of paroxysmal atrial fibrillation as per the hospital standard of care.

Exclusion Criteria:

* Persistent or Long standing AF
* CABG procedure within the last 180 days (six months).
* Documented left atrial thrombus on imaging [e.g. Transesophageal echocardiogram (TEE)].
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation (i.e. heparin or warfarin).
* Enrollment in another investigational study evaluating device or drug that might impact the results of this study.
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable).
* Acute illness or active systemic infection or sepsis.
* Life expectancy less than 12 months.
* Uncontrolled heart failure or NYHA class IV heart failure.
* Myocardial Infarction within 8 weeks of enrollment or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Procedural parameters | 6 months
  * Ablation parameters (such as average power delivered , average tip temperature , average impedance )
  * Lesion locations (such as PVI, Septal line, Mitral isthmus, CTI or any other lesion location)
  * Mapping techniques (Mapping system and catheter)
  * RF application time ( Calculated from the total number of RF application and duration of each RF application)
  * Ablation procedure time (Time from the first to the last RF application)
  * Total irrigation fluid administered during ablation procedure
  * Fluoroscopy time
AF Recurrence | 6 months
  * Recurrence of AF through six months post last RF ablation procedure using Cool Flex catheter. A 24 hour Holter will be provided to the patients for six month follow-up visit in order to monitor AF episodes. An AF episode will be considered a recurrence only if it lasts for 30 seconds or more.
  * AF recurrences during the blanking period (defined below) will not be reported.
Serious Adverse Events | 6 months
  All serious adverse events through six month follow-up

CONTACTS AND LOCATIONS:
Locations (6):
- Royal Adelaide Hospital, Adelaide, Australia
- Hopital du Haut Leveque, Pessac, France
- Universitat Leipzig Herzzentrum, Leipzig, Germany
- Ospendale dell'Angelo, Mestre, Italy
- Hospital Santa Cruz, Lisbon, Portugal
- Heart Hospital, London, United Kingdom